CLINICAL TRIAL: NCT02709525
Title: Use of Hyaluronic Acid as a Therapeutic Strategy for Bone Repair in Human: a Split-mouth Randomized Triple-blind Clinical Trial
Brief Title: Use of Hyaluronic Acid as a Therapeutic Strategy for Bone Repair in Human
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Carlos Eduardo Pinto de Alcântara, MSc,PhD Student, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 0328.0.203.000-10
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Alveolar Bone Loss
Keywords: hyaluronic acid; bone repair; dental socket; cone beam computed tomography
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hyaluronic acid (Experimental): Immediately after the extractions, one socket was randomly filled with 1% hyaluronic acid gel.
  Interventions: Drug: hyaluronic acid
- Blood clot (Placebo Comparator): Immediately after the extractions, the other side socket was naturally filled with blood clot.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: hyaluronic acid
  Other Names: Hyaluronan; Sodium hyaluronate
  Arms: hyaluronic acid
Other: Placebo
  Arms: Blood clot

SUMMARY:
The aim of this study is to evaluate the effects of hyaluronic acid (HA) on bone healing in human dental sockets.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic need for bilateral extraction of lower first premolars

Exclusion Criteria:

* Alcoholism, smoking, drug use and abuse of drugs; Systemic diseases: uncontrolled diabetes, blood dyscrasias, kidney or heart failure and osteoporosis; clinical or radiographic signs of pathological processes in the bone;

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of bone formation | 30 days after extraction and treatment application
  During the postoperative interval of 30 days, the patients underwent cone beam computed tomography (CBCT). Five central transverse scan images were captured from each socket. Using the KS300 software, the gray intensity was measured in each image and the results were expressed as mean percentage of bone formation
Fractal dimension | 30 days after extraction and treatment application
  During the postoperative interval of 30 days, the patients underwent cone beam computed tomography (CBCT). Five central transverse scan images were captured from each socket. The pattern of the alveolar trabecular bone was also evaluated through the fractal dimension in each image.
Dimensional Alveolar changes | 30 to 90 days after extraction and treatment application
  To determine whether treatment could prevent loss of buccolingual thickness, was compared bone loss of 90 to 30 days between the treated and control groups.
Percentage of bone formation | 90 days after extraction and treatment application
  During the postoperative interval of 90 days, the patients underwent cone beam computed tomography (CBCT). Five central transverse scan images were captured from each socket. Using the KS300 software, the gray intensity was measured in each image and the results were expressed as mean percentage of bone formation
Fractal dimension | 90 days after extraction and treatment application
  During the postoperative interval of 90 days, the patients underwent cone beam computed tomography (CBCT). Five central transverse scan images were captured from each socket. The pattern of the alveolar trabecular bone was also evaluated through the fractal dimension in each image.

CONTACTS AND LOCATIONS:
Overall Officials: Anderson Ferreira, Professor, Study Director — Instituto de Ciências Biológicas - Universidade Federal de Minas Gerais